CLINICAL TRIAL: NCT02780583
Title: Randomized Placebo Controlled Trial of Subcutaneous rhIL-1A (Anakinra) in the Management of Hospitalized Pediatric and Adult Patients With Macrophage Activation Syndrome
Brief Title: Treatment of Macrophage Activation Syndrome (MAS) With Anakinra
Acronym: MAS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: no further funding to continue, investigator relocated, no replacement found to continue
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, W Winn Chatham, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F151008003; FWA00005960 (Other Grant/Funding Number: DEPT. HEALTH AND HUMAN SERVICES); SOBI_UAB01 (Other Grant/Funding Number: Sweedish Orphan Biovitrum)
Record Dates: First submitted 2016-05-11; First posted 2016-05-23 (Estimated); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Macrophage Activation Syndrome
MeSH Terms: conditions — Macrophage Activation Syndrome | interventions — Interleukin 1 Receptor Antagonist Protein; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): methylprednisolone intravenously, placebo shots every 6 hours
  Interventions: Drug: placebo
- anakinra (Kineret) (Experimental): methylprednisolone intravenously, anakinra shots every 6 hours
  Interventions: Drug: kineret

INTERVENTIONS:
Drug: kineret — anakinra administered subcutaneously every 6 hours x 72 hours along with intravenous methylprednisolone
  Other Names: Anakinra
  Arms: anakinra (Kineret)
Drug: placebo — placebo injection administered every 6 hours along with intravenous methylprednisolone
  Other Names: normal saline
  Arms: placebo

SUMMARY:
The primary purpose of this study is to determine whether giving injections of anakinra is a safe and well tolerated treatment to give as an adjunct to standard prescribed treatment for patients who are admitted to the hospital with signs of severe inflammation (macrophage activation syndrome) that is potentially life-threatening. Anakinra is a commercially available product (Kineret™) approved for the treatment of rheumatoid arthritis; it is a replica of a naturally occurring protein called Il-1 receptor antagonist (IL-1ra), made by humans to inhibit and regulate the action of interleukin-1 (IL-1). IL-1 is a mediator of inflammation that when generated in excess amounts by immune system cells can result in severe dysfunction of multiple organs that can be life-threatening. The specific primary objectives of the study are to determine if giving anakinra results in no increased infection complications or mortality. Additional data will be collected to determine whether anakinra administration results in any other unanticipated side effects in this setting, and the effects of anakinra administration on inflammation markers, the overall dose of steroids required to treat the inflammation, and the length of hospital stay.

DETAILED DESCRIPTION:
Macrophage activation syndrome (MAS) is a disorder whereby the immune system generates very high levels of substances (cytokines) that promote inflammation to the extent dysfunction occurs in multiple organ systems which if unchecked, is frequently fatal to the affected individual. This can occur in the setting of a number of different immune system disorders including, systemic lupus, systemic-onset juvenile arthritis, and adult-onset Still's disease. MAS can also occur in response to infection with certain viruses such as Epstein-Barr virus (EBV) and malignancies involving lymphocytes.

Because of the high fatality of MAS (>50%), a number of different treatments have been tried to manage this disorder, including use of high-dose steroids, immune suppressants such as cyclosporine, and cytotoxic chemotherapy treatments (etoposide) with variable success and/or severe complications of immune suppression (as may occur with etoposide). A number of recent case reports and case series have reported success using cytokine-blocking therapies such as anakinra in the treatment of MAS that is associated with systemic-onset juvenile idiopathic arthritis and adult Still's disease. Anakinra is a bio-engineered form of the naturally occurring interleukin-1 receptor antagonist (IL-1ra), that blocks the action of interleukin-1, one of the cytokines that is expressed and present in very high amounts in patients who have MAS. Anakinra/Il-1ra is an attractive treatment for patients presenting with clinical features of MAS because it has a relatively short half-life and is easy to administer by subcutaneous injection. In previous trials of its use in patients with clinical features of bacterial sepsis (fever, elevated heart rate, low/falling blood pressure) , it was shown that anakinra does not have a harmful effect but also did not appear to have any benefit with repect to the defined primary outcome of improved survival. However, a recent re-analysis of the data accumulated in these same previous sepsis trials (for which the primary defined outcome was survival) indicates that survival was actually increased in the subgroup of sepsis patients with features of MAS (ferritin elevations in excess of 2,000 ng/ml, signs of coagulopathy, and liver enzyme elevations) who were randomized to receive anakinra compared to the subgroup of sepsis patients with features of MAS who were randomized to receive placebo.

Previous doses of anakinra up to 3500 mg/day over 72 hours that were employed in the trials of adult patients with sepsis were noted to be well tolerated without increased adverse outcomes compared to patients randomized to placebo. Recent case reports have shown that doses up to 100 mg every 6 hours were efficacious and well tolerated in children with systemic onset juvenile arthritis complicated by refractory macrophage activation syndrome.

This study will be the first controlled study to confirm whether anakinra at dose of 10 mg/kg/day to a maximum of dose of 200 mg/day divided every 12 hours (for children ≤40 kg) or 5 mg/kg/day up to a maximum dose of 400 mg/day divided every 6 hours (children > 40 kg and adults) does not result in increased mortality or infection complications when administered in addition to current UAB standard of care treatment (corticosteroids) to children and adults hospitalized with suspected macrophage activation syndrome.

ELIGIBILITY:
Inclusion Criteria:1] Previous diagnosis of systemic juvenile idiopathic arthritis (sJIA) and fulfills the Ravelli criteria (4) for macrophage activation syndrome with either:

two or more Laboratory criteria: 1. Decreased platelet count (≤262 ×10 9/L) 2. Elevated levels of aspartate aminotransferase (>59 U/L) 3. Decreased white blood cell count (≤4.0 × 109/L) 4. Hypofibrinogenemia (≤2.5 g/L) or, three or more combined clinical/laboratory criteria:

1. Decreased platelet count (≤262 × 109/L)
2. Elevated levels of aspartate aminotransferase (>59 U/L)
3. Decreased white blood cell count (≤4.0 × 109/L)
4. Hypofibrinogenemia (≤2.5 g/L)
5. Central nervous system dysfunction (irritability, disorientation, lethargy, seizures, coma)
6. Hemorrhages (purpura, easy bruising, mucosal bleeding)
7. Hepatomegaly (≥3 cm below the costal margin or confirmed by imaging)

OR

2] No previous diagnosis of sJIA and serum ferritin > 2,000 ng/ml and 3 out of the following:

1. Bicytopenia with two of the following:

   1. Absolute Neutrophil Count < 1,000,
   2. Platelets < 100, 000/mm3,
   3. Hemoglobin < 9 mg/dl
2. Fasting triglyceride >265 mg/dL
3. Splenomegaly
4. ALT OR AST > 120 IU/L (or > 2x upper limit of normal)
5. Fever with temp ≥ 101° F
6. Fibrinogen < 1.5 g/L (150 mg/dl) or INR > 1.5 or d-dimer > 500 ng/ml

   -

Exclusion Criteria:

1. Evidence of malignancy
2. Culture evidence of systemic bacterial infection at the time of screening
3. Known EBV viremia by PCR at time of screening (positive serologies are not an exclusion; results of EBV testing will not be necessary for enrollment, but may be ordered as part of the standard of care assessment to guide future management as results become available)
4. Previous treatment for the current MAS episode with corticosteroids, anakinra, tocilizumab, anti-TNF therapy or cyclosporine
5. <1 year of age
6. Family history of familial HLH
7. Evidence of any of the following

   1. Creatinine at the time of screening > 2X ULN or > twofold increase from patient's baseline creatinine within past 3 months (if known)
   2. Albumin < 1.5 at the time of screening
   3. Mechanical ventilation at the time of screening
   4. Hypotension requiring use of pressors at the time of screening

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Number of acquired infections, deaths in treatment group vs placebo group | within 72 hours after baseline
  The primary outcome measure is to determine whether hospital acquired infections or deaths are increased when anakinra is added to corticosteroid use during the first 72 hours of MAS management

SECONDARY OUTCOMES:
Normalization of elevations of MAS activity markers in treatment group vs placebo group | baseline to 72 hours after baseline
  Another purpose of this study is to determine whether adding anakinra to corticosteroids in the first 72 hours of MAS treatment results in greater normalization of MAS activity markers including serum ferritin, CRP, LDH, d-dimer/fibrinogen
Total corticosteroid use and chemotherapy rescue treatment in anakinra treated group vs placebo treated group | 2 years post enrollment
  Determine if treatment anakinra decreases the overall doses of steroids required to effectively manage anakinra, and if treatment with anakinra decreases the need to use chemotherapy drugs (etoposide) to treat MAS.

CONTACTS AND LOCATIONS:
Overall Officials: Walter W Chatham, MD, Principal Investigator — University of Alabama Hospital; Randall Q Cron, MD, Principal Investigator — Children's Hospital of Alabama
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Nurse Study Coordinators will gather and enter data
Supporting Information: Study Protocol, CSR
Time Frame: Dec 31 2020
Access Criteria: request to investigator

REFERENCES:
- [Derived] Cron RQ, Chatham WW. The Rheumatologist's Role in COVID-19. J Rheumatol. 2020 May 1;47(5):639-642. doi: 10.3899/jrheum.200334. Epub 2020 Mar 24. No abstract available. PMID 32209661
- [Derived] Eloseily EM, Weiser P, Crayne CB, Haines H, Mannion ML, Stoll ML, Beukelman T, Atkinson TP, Cron RQ. Benefit of Anakinra in Treating Pediatric Secondary Hemophagocytic Lymphohistiocytosis. Arthritis Rheumatol. 2020 Feb;72(2):326-334. doi: 10.1002/art.41103. Epub 2019 Dec 26. PMID 31513353